CLINICAL TRIAL: NCT03128606
Title: Assessment of Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG3067, the Combination of GLPG3067 and GLPG2222, and the Combination of GLPG3067, GLPG2222 and GLPG2737 in Healthy Female Subjects, Including a Relative Bioavailability and Food Effect Part for Single Dose of GLPG3067.
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of GLPG3067 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3067-CL-101
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (13):
- GLPG3067 single dose (Experimental): Single dose of GLPG3067 oral suspension at up to 6 dose levels in ascending order.
  Interventions: Drug: GLPG3067 single dose
- Placebo single dose (Placebo Comparator): Single dose of Placebo oral suspension.
  Interventions: Drug: Placebo single dose
- GLPG3067 oral suspension fed 1 (Experimental): Single dose 1 of GLPG3067 oral suspension after a standardized breakfast.
  Interventions: Drug: GLPG3067 oral suspension
- GLPG3067 oral tablet fed 1 (Experimental): Single dose 1 of GLPG3067 oral tablet after a standardized breakfast.
  Interventions: Drug: GLPG3067 oral tablet
- GLPG3067 oral tablet fasted 1 (Experimental): Single dose 1 of GLPG3067 oral tablet after an overnight fast.
  Interventions: Drug: GLPG3067 oral tablet
- GLPG3067 oral tablet fed 2 (Experimental): Single dose 2 of GLPG3067 oral tablet after a standardized breakfast.
  Interventions: Drug: GLPG3067 oral tablet
- GLPG3067 oral tablet fed 2 high-fat high-calorie (Experimental): Single dose 2 of GLPG3067 oral tablet after a high-fat high-calorie breakfast
  Interventions: Drug: GLPG3067 oral tablet
- GLPG3067 multiple dose (Experimental): Multiple doses of GLPG3067 oral suspension at up to 5 dose levels in ascending order.
  Interventions: Drug: GLPG3067 multiple dose
- Placebo multiple dose (Placebo Comparator): Multiple doses of Placebo oral suspension.
  Interventions: Drug: Placebo multiple dose
- GLPG3067/GLPG2222 multiple dose (Experimental): Multiple doses of GLPG3067 oral suspension combined with GLPG2222 oral tablet up to 2 dose levels in ascending order.
  Interventions: Drug: GLPG3067/GLPG2222 multiple dose
- GLPG3067/GLPG2222 Placebo multiple dose (Placebo Comparator): Multiple doses of GLPG3067 matching placebo oral suspension combined with GLPG2222 matching placebo oral tablet.
  Interventions: Drug: GLPG3067/GLPG2222 Placebo multiple dose
- GLPG3067/GLPG2222/GLPG2737 multiple dose (Experimental): Multiple doses of GLPG3067 oral tablet combined with GLPG2222 oral tablet and GLPG2737 oral capsule at up to 2 dose levels in ascending order.
  Interventions: Drug: GLPG3067/GLPG2222/GLPG2737 multiple dose
- GLPG3067/GLPG2222/GLPG2737 Placebo multiple dose (Placebo Comparator): Multiple doses of GLPG3067 matching placebo oral tablet combined with GLPG2222 matching placebo oral tablet and GLPG2737 matching placebo oral capsule.
  Interventions: Drug: GLPG3067/GLPG2222/GLPG2737 Placebo multiple dose

INTERVENTIONS:
Drug: GLPG3067 single dose — GLPG3067 oral suspension, single ascending doses, daily
  Arms: GLPG3067 single dose
Drug: Placebo single dose — Placebo, oral suspension, daily
  Arms: Placebo single dose
Drug: GLPG3067 multiple dose — GLPG3067 oral suspension, multiple ascending doses, daily for 14 days
  Arms: GLPG3067 multiple dose
Drug: Placebo multiple dose — Placebo, oral suspension, daily for 14 days
  Arms: Placebo multiple dose
Drug: GLPG3067 oral suspension — GLPG3067 oral suspension, single dose, daily
  Arms: GLPG3067 oral suspension fed 1
Drug: GLPG3067 oral tablet — GLPG3067 oral tablet, single dose, daily
  Arms: GLPG3067 oral tablet fasted 1; GLPG3067 oral tablet fed 1; GLPG3067 oral tablet fed 2; GLPG3067 oral tablet fed 2 high-fat high-calorie
Drug: GLPG3067/GLPG2222 multiple dose — GLPG3067 oral suspension and GLPG2222 oral tablet, multiple doses, daily for 14 days
  Arms: GLPG3067/GLPG2222 multiple dose
Drug: GLPG3067/GLPG2222 Placebo multiple dose — GLPG3067 matching placebo oral suspension and GLPG2222 matching placebo oral tablet, multiple doses, daily for 14 days
  Arms: GLPG3067/GLPG2222 Placebo multiple dose
Drug: GLPG3067/GLPG2222/GLPG2737 multiple dose — GLPG3067 oral tablet, GLPG2222 oral tablet and GLPG2737 oral capsule, multiple doses, daily for 14 days
  Arms: GLPG3067/GLPG2222/GLPG2737 multiple dose
Drug: GLPG3067/GLPG2222/GLPG2737 Placebo multiple dose — GLPG3067 matching placebo oral tablet, GLPG2222 matching placebo oral tablet and GLPG2737 matching placebo oral capsule, multiple doses, daily for 14 days
  Arms: GLPG3067/GLPG2222/GLPG2737 Placebo multiple dose

SUMMARY:
The study is a First-in-Human, Phase I, randomized, double-blind, placebo-controlled, single center study, evaluating single and multiple ascending oral doses of GLPG3067 and the combination of GLPG3067 and GLPG2222 and the combination of GLPG3067,GLPG2222 and GLPG2737 given for 14 days in healthy women of non-childbearing potential.

The purpose of the study is to evaluate the safety and tolerability of single ascending oral doses and multiple ascending oral doses of GLPG3067 given to healthy women of non-childbearing potential compared to placebo, as well as of multiple oral doses of the combination of GLPG3067/GLPG2222 compared to matching placebo for each compound and multiple oral doses of the combination of GLPG3067/GLPG2222/GLPG2737 compared to matching placebo for each compound.

ELIGIBILITY:
Inclusion Criteria:

* Female subject between 18-70 years of age, inclusive, on the date of signing the informed consent form (ICF).
* Be of non-childbearing potential defined as surgically sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy), or post-menopausal (at least 12 consecutive months without menstruation, without an alternative medical cause [including hormone replacement therapy]).
* Have a body mass index between 18-30 kg/m2, inclusive.
* Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead triplicate electrocardiogram (ECG), and clinical safety laboratory tests prior to the initial study drug administration.
* Discontinuation of all medications (including over-the-counter and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements, and hormonal replacement therapy for postmenopausal subjects) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) at least 2 weeks prior to the first study drug administration.

Exclusion Criteria:

* Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
* Clinically significant symptoms or illness in the 3 months before screening.
* Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Any laboratory result considered by the investigator as clinically significant prior to study drug administration.
* Creatinine clearance ≤80 mL/min using the Cockcroft-Gault formula for subjects aged ≤50 years, or creatinine clearance ≤70 mL/min using the Cockcroft-Gault formula for subjects aged >50 years. A 24-hour urine collection to determine the actual value may be performed to confirm creatinine clearance if required.
* Clinically significant abnormalities of vital signs at screening.
* Clinically relevant abnormalities detected on ECG regarding either rhythm or conduction (e.g. QT interval corrected for heart rate using Fridericia's formula [QTcF] >470 ms) or a known long QT syndrome. A first degree heart block or sinus arrhythmia will not be considered as a significant abnormality.
* Participation in a drug, drug and device delivery system or combination, or biologic investigational research study within 8 weeks or 5 times the half-life of the investigational drug, if the half-life is known (whichever is longer) prior to initial study drug administration. Subjects who have been dosed previously with GLPG3067 in a clinical trial are allowed to participate Part 4 of this study as long as they completed their last follow-up visit or a washout period of 5 times the half-life of GLPG3067 (whichever is longer) after the last study drug administration is respected.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Change versus placebo in the proportion of subjects with adverse events | Between screening and 14 days after the last dose
  To assess safety and tolerability of single ascending doses, multiple ascending doses of GLPG3067 alone, or in combination with GLPG2222, or in combination with GLPG2222 and GLPG2737 versus placebo in healthy subjects

SECONDARY OUTCOMES:
Maximum observed plasma concentration of GLPG3067 (Cmax) given alone or in combination with GLPG2222 or in combination with GLPG2222 and GLPG2737 | Between Day 1 predose and 10 days after the last dose
  To characterize pharmacokinetics of GLPG3067 after a single oral dose and of GLPG3067, GLPG2222, and GLPG2737 after multiple oral doses in healthy subjects
Area under the plasma concentration-time curve of GLPG3067 (AUC0-t) given alone or in combination with GLPG2222 or in combination with GLPG2222 and GLPG2737 | Between Day 1 predose and 10 days after the last dose
  To characterize pharmacokinetics of GLPG3067 after a single oral dose and of GLPG3067, GLPG2222, and GLPG2737 after multiple oral doses in healthy subjects
Ratio of 4-beta-hydroxycholesterol/cholesterol in plasma after multiple oral doses in healthy subjects | Day 1 predose and Day 14
  To assess the potential for CYP3A4 interaction with GLPG3067, GLPG3067 and GLPG2222, or GLPG3067 and GLPG2222 and GLPG2737
Maximum observed plasma concentration of GLPG3067 (Cmax) given alone in fed state | Between Day 1 predose and 10 days after the last dose
  To assess the relative bioavailability of GLPG3067 when given as a single dose of oral suspension or an oral tablet both administered in fed state
Concentration in plasma observed at 24 hours post dose (C24h) of GLPG3067 given alone in fed state | Between Day 1 predose and 10 days after the last dose
  To assess the relative bioavailability of GLPG3067 when given as a single dose of oral suspension or an oral tablet both administered in fed state
Area under the plasma concentration-time curve of GLPG3067 (AUC0-t) given alone in fed state | Between Day 1 predose and 10 days after the last dose
  To assess the relative bioavailability of GLPG3067 when given as a single dose of oral suspension or an oral tablet both administered in fed state
Maximum observed plasma concentration of GLPG3067 (Cmax) given alone in fasted state | Between Day 1 predose and 10 days after the last dose
  To assess the effect of food on the pharmacokinetics of GLPG3067 when given under fasted versus fed conditions
Concentration in plasma observed at 24 hours post dose (C24h) of GLPG3067 given alone in fasted state | Between Day 1 predose and 10 days after the last dose
  To assess the effect of food on the pharmacokinetics of GLPG3067 when given under fasted versus fed conditions
Area under the plasma concentration-time curve of GLPG3067 (AUC0-t) given alone in fasted state | Between Day 1 predose and 10 days after the last dose
  To assess the effect of food on the pharmacokinetics of GLPG3067 when given under fasted versus fed conditions

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided